CLINICAL TRIAL: NCT01108796
Title: Additional Effect of a Life Style Program on Antihypertensive Treatment With Telmisartan
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.579
Record Dates: First submitted 2010-03-11; First posted 2010-04-22 (Estimated); Results first posted 2011-12-30 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients at cardiovascular risk

SUMMARY:
This post-marketing surveillance study is designed to supplement the data on efficacy and tolerability of Micardis® and MicardisPlus® in patients at cardiovascular risk under general practice conditions.

The aim of the study is to investigate the effect of a six-month treatment with Micardis® / MicardisPlus® on blood pressure and the effect of the Lifestyle education tool for weight reduction on blood pressure control.

In addition, the post-marketing surveillance study will provide information on the effects on target measurement of the Lifestyle education tool and various laboratory parameters produced by treatment with Micardis® and MicardisPlus® in an unselected patient population under general practice conditions.

ELIGIBILITY:
Inclusion criteria:

1. Patients with essential hypertension (blood pressure (BP) higher or equal to 140/90 mmHg or higher or equal to 130/80 mmHg in case of diabetic patients)
2. Patients with hypertension under treatment with one or more antihypertensive drug

Exclusion criteria:

Patients are excluded according to the summary of product characteristics (SmPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypertension
Sampling Method: Probability Sample
Enrollment: 1856 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (182):
- Slovenia (182):
  - Boehringer Ingelheim Investigational Site 34, ?adca
  - Boehringer Ingelheim Investigational Site 2, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 3, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 4, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 5, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 6, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 7, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 8, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 10, Bardejov
  - Boehringer Ingelheim Investigational Site 11, Bardejov
  - Boehringer Ingelheim Investigational Site 12, Bardejov
  - Boehringer Ingelheim Investigational Site 9, Bardejov
  - Boehringer Ingelheim Investigational Site 1, Bánovce Nad Bebravou
  - Boehringer Ingelheim Investigational Site 13, Bratislava
  - Boehringer Ingelheim Investigational Site 14, Bratislava
  - Boehringer Ingelheim Investigational Site 15, Bratislava
  - Boehringer Ingelheim Investigational Site 16, Bratislava
  - Boehringer Ingelheim Investigational Site 17, Bratislava
  - Boehringer Ingelheim Investigational Site 18, Bratislava
  - Boehringer Ingelheim Investigational Site 19, Bratislava
  - Boehringer Ingelheim Investigational Site 20, Bratislava
  - Boehringer Ingelheim Investigational Site 21, Bratislava
  - Boehringer Ingelheim Investigational Site 22, Bratislava
  - Boehringer Ingelheim Investigational Site 23, Bratislava
  - Boehringer Ingelheim Investigational Site 24, Bratislava
  - Boehringer Ingelheim Investigational Site 25, Bratislava
  - Boehringer Ingelheim Investigational Site 26, Bratislava
  - Boehringer Ingelheim Investigational Site 27, Bratislava
  - Boehringer Ingelheim Investigational Site 28, Bratislava
  - Boehringer Ingelheim Investigational Site 29, Brezno
  - Boehringer Ingelheim Investigational Site 30, Brezno
  - Boehringer Ingelheim Investigational Site 31, Brezno
  - Boehringer Ingelheim Investigational Site 32, Brezno
  - Boehringer Ingelheim Investigational Site 33, Byt?a
  - Boehringer Ingelheim Investigational Site 35, Dolný Kubín
  - Boehringer Ingelheim Investigational Site 36, Dubnica Nad Váhom
  - Boehringer Ingelheim Investigational Site 37, Dubnica Nad Váhom
  - Boehringer Ingelheim Investigational Site 38, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 39, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 40, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 41, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 42, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 43, Dunajská Streda
  - Boehringer Ingelheim Investigational Site 44, Galanta
  - Boehringer Ingelheim Investigational Site 45, Galanta
  - Boehringer Ingelheim Investigational Site 46, Handlová
  - Boehringer Ingelheim Investigational Site 47, Hlohovec
  - Boehringer Ingelheim Investigational Site 48, Hlohovec
  - Boehringer Ingelheim Investigational Site 49, Hnús?a
  - Boehringer Ingelheim Investigational Site 50, Hurbanovo
  - Boehringer Ingelheim Investigational Site 51, Jesenské
  - Boehringer Ingelheim Investigational Site 52, Kezmarok
  - Boehringer Ingelheim Investigational Site 53, Kolárovo
  - Boehringer Ingelheim Investigational Site 54, Komárno
  - Boehringer Ingelheim Investigational Site 55, Komárno
  - Boehringer Ingelheim Investigational Site 56, Kosice
  - Boehringer Ingelheim Investigational Site 57, Kosice
  - Boehringer Ingelheim Investigational Site 58, Kosice
  - Boehringer Ingelheim Investigational Site 59, Kosice
  - Boehringer Ingelheim Investigational Site 60, Kosice
  - Boehringer Ingelheim Investigational Site 61, Kosice
  - Boehringer Ingelheim Investigational Site 62, Kosice
  - Boehringer Ingelheim Investigational Site 63, Kosice
  - Boehringer Ingelheim Investigational Site 64, Kosice
  - Boehringer Ingelheim Investigational Site 65, Kosice
  - Boehringer Ingelheim Investigational Site 66, Kosice
  - Boehringer Ingelheim Investigational Site 67, Kosice
  - Boehringer Ingelheim Investigational Site 68, Kosice
  - Boehringer Ingelheim Investigational Site 69, Kosice
  - Boehringer Ingelheim Investigational Site 70, Kosice
  - Boehringer Ingelheim Investigational Site 71, Krá?ovský Chlmec
  - Boehringer Ingelheim Investigational Site 72, Kysucké Nové Mesto
  - Boehringer Ingelheim Investigational Site 73, Kysucké Nové Mesto
  - Boehringer Ingelheim Investigational Site 74, Kysucké Nové Mesto
  - Boehringer Ingelheim Investigational Site 75, Levice
  - Boehringer Ingelheim Investigational Site 76, Levice
  - Boehringer Ingelheim Investigational Site 77, Levice
  - Boehringer Ingelheim Investigational Site 78, Lipany
  - Boehringer Ingelheim Investigational Site 79, Lu?enec
  - Boehringer Ingelheim Investigational Site 80, Lu?enec
  - Boehringer Ingelheim Investigational Site 81, Lu?enec
  - Boehringer Ingelheim Investigational Site 82, Lu?enec
  - Boehringer Ingelheim Investigational Site 83, Martin
  - Boehringer Ingelheim Investigational Site 84, Martin
  - Boehringer Ingelheim Investigational Site 85, Martin
  - Boehringer Ingelheim Investigational Site 86, Michalovce
  - Boehringer Ingelheim Investigational Site 87, Michalovce
  - Boehringer Ingelheim Investigational Site 88, Michalovce
  - Boehringer Ingelheim Investigational Site 89, Myjava
  - Boehringer Ingelheim Investigational Site 90, Námestovo
  - Boehringer Ingelheim Investigational Site 91, Nitra
  - Boehringer Ingelheim Investigational Site 92, Nitra
  - Boehringer Ingelheim Investigational Site 93, Nitra
  - Boehringer Ingelheim Investigational Site 94, Nitra
  - Boehringer Ingelheim Investigational Site 95, Nové Mesto Nad Váhom
  - Boehringer Ingelheim Investigational Site 96, Nové Mesto Nad Váhom
  - Boehringer Ingelheim Investigational Site 97, Nové Mesto Nad Váhom
  - Boehringer Ingelheim Investigational Site 100, Nové Zámky
  - Boehringer Ingelheim Investigational Site 101, Nové Zámky
  - Boehringer Ingelheim Investigational Site 98, Nové Zámky
  - Boehringer Ingelheim Investigational Site 99, Nové Zámky
  - Boehringer Ingelheim Investigational Site 102, Partizánske
  - Boehringer Ingelheim Investigational Site 103, Partizánske
  - Boehringer Ingelheim Investigational Site 104, Pezinok
  - Boehringer Ingelheim Investigational Site 105, Pies?any
  - Boehringer Ingelheim Investigational Site 106, Poprad
  - Boehringer Ingelheim Investigational Site 107, Poprad
  - Boehringer Ingelheim Investigational Site 108, Poprad
  - Boehringer Ingelheim Investigational Site 109, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 110, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 111, Presov
  - Boehringer Ingelheim Investigational Site 112, Presov
  - Boehringer Ingelheim Investigational Site 113, Presov
  - Boehringer Ingelheim Investigational Site 114, Presov
  - Boehringer Ingelheim Investigational Site 115, Prievidza
  - Boehringer Ingelheim Investigational Site 116, Prievidza
  - Boehringer Ingelheim Investigational Site 117, Prievidza
  - Boehringer Ingelheim Investigational Site 118, Rajec
  - Boehringer Ingelheim Investigational Site 119, Revúca
  - Boehringer Ingelheim Investigational Site 120, Revúca
  - Boehringer Ingelheim Investigational Site 121, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 122, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 123, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 124, Roz?ava
  - Boehringer Ingelheim Investigational Site 125, Roz?ava
  - Boehringer Ingelheim Investigational Site 126, Ruzomberok
  - Boehringer Ingelheim Investigational Site 127, Ruzomberok
  - Boehringer Ingelheim Investigational Site 128, Sa?a
  - Boehringer Ingelheim Investigational Site 129, Sa?a
  - Boehringer Ingelheim Investigational Site 130, Sa?a
  - Boehringer Ingelheim Investigational Site 131, Se?ovce
  - Boehringer Ingelheim Investigational Site 132, Se?ovce
  - Boehringer Ingelheim Investigational Site 133, Skalica
  - Boehringer Ingelheim Investigational Site 134, Snina
  - Boehringer Ingelheim Investigational Site 135, Snina
  - Boehringer Ingelheim Investigational Site 136, Spisská Nová Ves
  - Boehringer Ingelheim Investigational Site 137, Spisská Nová Ves
  - Boehringer Ingelheim Investigational Site 138, Stará ?ubov?a
  - Boehringer Ingelheim Investigational Site 139, Stará ?ubov?a
  - Boehringer Ingelheim Investigational Site 140, Stará ?ubov?a
  - Boehringer Ingelheim Investigational Site 141, Stropkov
  - Boehringer Ingelheim Investigational Site 142, Stúrovo
  - Boehringer Ingelheim Investigational Site 143, Surany
  - Boehringer Ingelheim Investigational Site 144, Surany
  - Boehringer Ingelheim Investigational Site 145, Svit
  - Boehringer Ingelheim Investigational Site 146, Topo??any
  - Boehringer Ingelheim Investigational Site 147, Torna?a
  - Boehringer Ingelheim Investigational Site 148, Trebisov
  - Boehringer Ingelheim Investigational Site 149, Trebisov
  - Boehringer Ingelheim Investigational Site 150, Trebisov
  - Boehringer Ingelheim Investigational Site 151, Tren?ín
  - Boehringer Ingelheim Investigational Site 152, Tren?ín
  - Boehringer Ingelheim Investigational Site 153, Tren?ín
  - Boehringer Ingelheim Investigational Site 154, Tren?ín
  - Boehringer Ingelheim Investigational Site 155, Trnava
  - Boehringer Ingelheim Investigational Site 156, Trnava
  - Boehringer Ingelheim Investigational Site 157, Trnava
  - Boehringer Ingelheim Investigational Site 158, Trnava
  - Boehringer Ingelheim Investigational Site 159, Trstená
  - Boehringer Ingelheim Investigational Site 160, Tur?ianske Teplice
  - Boehringer Ingelheim Investigational Site 161, Turzovka
  - Boehringer Ingelheim Investigational Site 162, Ve?ké Kapusany
  - Boehringer Ingelheim Investigational Site 163, Ve?ké Kapusany
  - Boehringer Ingelheim Investigational Site 164, Ve?ký Krtís
  - Boehringer Ingelheim Investigational Site 165, Ve?ký Krtís
  - Boehringer Ingelheim Investigational Site 167, Vranov Nad Top?ou
  - Boehringer Ingelheim Investigational Site 166, Vráble
  - Boehringer Ingelheim Investigational Site 168, Zarnovica
  - Boehringer Ingelheim Investigational Site 169, Zeliezovce
  - Boehringer Ingelheim Investigational Site 170, Zilina
  - Boehringer Ingelheim Investigational Site 171, Zilina
  - Boehringer Ingelheim Investigational Site 172, Zilina
  - Boehringer Ingelheim Investigational Site 173, Zilina
  - Boehringer Ingelheim Investigational Site 174, Zilina
  - Boehringer Ingelheim Investigational Site 175, Zilina
  - Boehringer Ingelheim Investigational Site 176, Zlaté Moravce
  - Boehringer Ingelheim Investigational Site 177, Zlaté Moravce
  - Boehringer Ingelheim Investigational Site 178, Zlaté Moravce
  - Boehringer Ingelheim Investigational Site 179, Zvolen
  - Boehringer Ingelheim Investigational Site 180, Zvolen
  - Boehringer Ingelheim Investigational Site 181, Zvolen
  - Boehringer Ingelheim Investigational Site 182, Zvolen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The aim of the study is to investigate the effect of the Lifestyle education tool (Tool/No Tool) for weight reduction on blood pressure control during a six-month treatment with Micardis® / MicardisPlus®. Patients were designated to participate or not participate in a Lifestyle education tool by the investigator under general practice conditions.
Pre-assignment Details: A total of 1856 were entered into this trial and 1841 were analysed. For 15 patients case report forms were not available or not usable for analysis
Groups:
- Micardis® (Telmisartan); MicardisPlus® (Telmisartan Hydrochlorothiazide): These patients in addition received Tool or No Tool treatment
Period: Overall Study
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide)
Started | 774 | 1067
Completed | 767 | 1060
Not Completed | 7 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Micardis® (Telmisartan): Patients were enrolled into two groups, receiving treatment with Micardis or MicardisPlus and in addition with Tool or No Tool. The system summarizes the number of patients automatically. The total number is always 1841.
- Total: Total of all reporting groups
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction) | Total
Number analyzed (Participants) | 774 | 1067 | 1187 | 654 | 3682
Age, Continuous [Mean (Standard Deviation); unit: Years] — Patients were enrolled into two groups, receiving treatment with Micardis or MicardisPlus and in addition with Tool or No Tool. The system summarizes the number of patients automatically. The total number is always 1841.
  Years | NA (NA) — Mean and Standard Deviation numbers of patients' age per Micardis®/Micardis Plus® arms not available in the statistical analysis report | NA (NA) — Mean and Standard Deviation numbers of patients' age per Micardis®/Micardis Plus® arms not available in the statistical analysis report | 61.14 (10.09) | 61.94 (11.01) | 61.43 (10.43)
Sex/Gender, Customized [Number; unit: Participants] — Patients were enrolled into two groups, receiving treatment with Micardis or MicardisPlus and in addition with Tool or No Tool. The system summarizes the number of patients automatically. The total number is always 1841.
  Participants
    Female, Tool/No Tool | 0 | 0 | 679 | 390 | 1069
    Male, Tool/No Tool | 0 | 0 | 507 | 264 | 771
    Female, Micardis®/MicardisPlus® | 445 | 624 | 0 | 0 | 1069
    Male, Micardis®/MicardisPlus® | 328 | 443 | 0 | 0 | 771

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mean Blood Pressure (Systolic) After Treatment, Compared to Baseline
Description: Changes in blood pressure in patients with systolic values, measured at baseline and final visit, by treatment and by Tool/No Tool
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 711 | 966 | 1083 | 594
mmHg | -30.71 (17.81) | -30.32 (15.05) | -30.35 (16.11) | -30.73 (16.58)

2. Primary Outcome: Changes in Mean Blood Pressure (Diastolic) After Treatment, Compared to Baseline
Description: Changes in blood pressure in patients with diastolic values, measured at baseline and final visit, by treatment and by Tool/No Tool
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 711 | 966 | 1083 | 594
mmHg | -14.73 (8.75) | -15.31 (8.87) | -15.29 (8.85) | -14.65 (8.76)

3. Secondary Outcome: Changes in Laboratory Parameters:Low Density Lipoprotein (LDL)
Description: Changes in LDL cholesterol levels from baseline to final visit in patients with both laboratory values valid, by treatment and by Tool/No Tool
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 434 | 577 | 709 | 302
mmol/l | -0.41 (0.65) | -0.51 (0.77) | -0.50 (0.74) | -0.40 (0.68)

4. Secondary Outcome: Changes in Laboratory Parameters:High Density Lipoprotein (HDL)
Description: as for outcome 3
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 441 | 571 | 714 | 298
mmol/l | 0.11 (0.25) | 0.09 (0.49) | 0.12 (0.31) | 0.06 (0.56)

5. Secondary Outcome: Changes in Laboratory Parameters: Triglycerides
Description: Changes in the triglyceride levels from baseline to final visit in patients with both laboratory values valid, by treatment and by Tool/No Tool
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 450 | 587 | 727 | 310
mmol/l | -0.24 (0.61) | -0.30 (0.80) | -0.32 (0.74) | -0.18 (0.69)

6. Secondary Outcome: Changes in Laboratory Parameters: Blood Glucose
Description: Changes in the fasting blood glucose levels from baseline to final visit in patients with both laboratory values valid, by treatment and by Tool/No Tool
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 457 | 595 | 746 | 306
mmol/l | -0.49 (1.19) | -0.45 (1.09) | -0.49 (1.17) | -0.42 (1.04)

7. Secondary Outcome: Assessment of Metabolic Effect
Description: Metabolic effect was rated by the investigators as 'positive', 'neutral' and 'negative'
Time Frame: 24 weeks (Visit 1 to Visit 3)
Measure: Number; unit: Participants
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide) | Tool (With Lifestyle Education Tool on Weight Reduction) | No Tool (Without Lifestyle Education Tool on Weight Reduction)
Number analyzed (Participants) | 774 | 1067 | 1187 | 654
Participants
  Positive | 544 | 695 | 835 | 404
  Neutral | 222 | 361 | 339 | 244
  Negative | 1 | 6 | 3 | 4
  Not available | 7 | 5 | 10 | 2

ADVERSE EVENTS:
Time Frame: 24 weeks/ 6 months
Arm/Group | Micardis® (Telmisartan) | MicardisPlus® (Telmisartan Hydrochlorothiazide)
Serious Adverse Events (participants affected / at risk) | 0/774 | 1/1067
Other Adverse Events (participants affected / at risk) | 0/774 | 0/1067
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micardis® (Telmisartan) (N=774) | MicardisPlus® (Telmisartan Hydrochlorothiazide) (N=1067)
Cerebrovascular accident (fatal stroke) (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract